CLINICAL TRIAL: NCT03685097
Title: Comparison of Two Point-of-care Devices for Viscoelastic Hemostasis Assays
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Collaborators: IRCCS Policlinico S. Donato (Other)
Responsible Party: Sponsor
Other Study IDs: HEMCS-013
Record Dates: First submitted 2018-09-21; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Cardiac surgery patients: Patients undergoing elective cardiac surgery requiring cardiopulmonary bypass.
  Interventions: Diagnostic Test: Quantra System with the QPlus Cartridge

INTERVENTIONS:
Diagnostic Test: Quantra System with the QPlus Cartridge — Point-of-care viscoelastic testing

SUMMARY:
This study will investigate the correlation and agreement of Quantra-derived parameters with parameters reported by the ROTEM delta and standard laboratory tests in cardiac surgery patients. In addition the association of Quantra-derived parameters with select platelet function tests will be investigated.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The Quantra QPlus Cartridge (previously called the Surgical Cartridge), was developed to monitor hemostasis during major surgical procedures in adult patients. The cartridge provides six parameters that depict the functional status of a patient's coagulation system.

This single site, prospective observational study will investigate the correlation and agreement of Quantra-derived parameters with parameters reported by the ROTEM delta and standard laboratory tests (PT, aPTT, fibrinogen, platelet count) in cardiac surgery patients. As an additional exploratory study, the association of Quantra-derived parameters with select platelet function tests will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years
* Subject is undergoing elective cardiac surgery with cardiopulmonary bypass
* Subject is willing to participate and has signed a consent form

Exclusion Criteria:

* Subject is younger than 18 years
* Subject has known congenital coagulopathy
* Subject is unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects 18 years or older undergoing cardiac surgery with cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Comparison of QPlus Clot Time and Clot Stiffness results to comparable ROTEM delta results | Baseline (before surgery)
  Coagulation function assessed by Quantra QPlus Cartridge and ROTEM delta
Comparison of QPlus Clot Time and Clot Stiffness results to comparable ROTEM delta | After cardiac bypass (10 minutes after administration of protamine)
  Coagulation function assessed by Quantra QPlus Cartridge and ROTEM delta
Comparison of QPlus Clot Time and Clot Stiffness results to standard coagulation test results | Baseline (before surgery)
  Coagulation function assessed by Quantra QPlus Cartridge and standard coagulation tests
Comparison of QPlus Clot Time and Clot Stiffness results to standard coagulation test results | After cardiac bypass (10 minutes after administration of protamine)
  Coagulation function assessed by Quantra QPlus Cartridge and standard coagulation tests

SECONDARY OUTCOMES:
Comparison of QPlus Clot Stiffness results to platelet function tests with multiple electrode aggregometry (MEA): ADPtest and TRAPtest | Baseline (before surgery)
  Platelet function assessed by Quantra QPlus Cartridge and MEA
Comparison of QPlus Clot Stiffness results to platelet function tests with multiple electrode aggregometry (MEA): ADPtest and TRAPtest | After cardiac bypass (10 minutes after administration of protamine)
  Platelet function assessed by Quantra QPlus Cartridge and MEA

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico San Donato (Milan) Italy
Locations (1):
- IRCCS Policlinico San Donato, Milan, Italy

IPD SHARING:
Plan to Share IPD: No